CLINICAL TRIAL: NCT04665219
Title: Health Belief Model for Empowering Parental Toothbrushing and Sugar Intake Control in Reducing Early Childhood Caries Among Young Children - a Cluster Randomized Controlled Trial
Brief Title: HBM for Empowering Parental Toothbrushing and Sugar Intake Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor May C.M. Wong, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HMRF (Ref: 17181971)
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Health Behavior; Mobile Phone Use; Early Childhood Caries
Keywords: Health Belief Model; Mobile Health; Early Childhood Caries; Oral Health Promotion
MeSH Terms: conditions — Health Behavior; Cell Phone Use

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Only receive a standard message.
  Interventions: Behavioral: Standard text message
- Test group (Experimental): Receive HBM-based messages.
  Interventions: Behavioral: HBM-based text messages

INTERVENTIONS:
Behavioral: HBM-based text messages — The intervention in the test group will consist of a set of text messages developed based on the HBM to be sent to the parents regularly in the following 48 weeks.
  During the first 24 weeks, parents will receive a text message (and feedback if deemed appropriate) each week. In the next 24 weeks, the parents will receive a text message every 4 weeks, altogether 30 messages will be sent to the parents. All messages will be sent to the parents individually through free mobile App by a research assistant.
  Arms: Test group
Behavioral: Standard text message — Parents in the control group will receive an oral health education pamphlet produced by the Oral Health Education Division in the Department of Health, the Government of Hong Kong SAR. In order to maintain a double-blind design in the present study, the pamphlet will be distributed in an electronic form and sent via a text message.
  Arms: Control group

SUMMARY:
It has been recognized that oral health education for parents is critical for the prevention of early childhood caries (ECC). Few parents practiced caries prevention procedures for their children in daily life, though. Inspired by Health Belief Model (HBM) and using text messaging as a vehicle, a novel intervention scheme will be developed in this study. The objective of the present randomized clinical trial (RCT) is to investigate the effectiveness of the HBM-based behavioral intervention using text message to reduce early childhood caries of children at age 4 through promoting the parental oral health care behaviors (toothbrushing and sugar intake control) for their young children compared to conventional oral health education. This RCT will recruit child-parent dyads in 26-36 child help centers or kindergartens with nursery classes located in Hong Kong. A total of 518-628 dyads will be recruited and randomly allocated into the test or control group with a 1:1 ratio. For parents in the test group, the intervention will consist of a set of HBM-based text messages sent regularly in the following 48 weeks. A standard text message will be sent to the parents in the control group. The primary outcome will be dental caries measured by dmft/dmfs of the children at 4 years old.

By HBM-based intervention via a low-cost text messaging vehicle, it should be able to help the parents establish proper oral health behaviors for their children and safeguard the oral health of children in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* young child aged18-30 months
* young children not having any severe medical conditions complicating oral health and dental examination
* parents having a mobile phone with certain Apps to receive the text messages in time (e.g. WhatsApp or WeChat)
* parents who can read Chinese

Exclusion Criteria:

* families that have been participating in another oral health promotion program

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 518 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
dmft/dmfs scores of the children at 4 years old | The children will be examined at the 24 months follow up. The tooth status of the erupted primary teeth would be assessed by careful visual inspection.
  The dental caries measured by dmft/dmfs (number of teeth/surfaces that are decayed missing or filled) of the children at aged 4 years (42-54 months).

SECONDARY OUTCOMES:
average frequency of parental toothbrushing per day | 24 months
  Change in parental oral health behavior over the study period, 2 times as preferred
average frequency of intake of sugary snack/drink per day | 24 months
  Change in parental oral health behavior over the study period, 2 times or less frequent as preferred
oral hygiene status using the Visible Plaque Index | 24 months
  The change in presence or absence of plaque on the buccal and lingual surfaces of all primary teeth over the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang K, Lee GHM, Liu P, Wong HC, Gao X, Wong SYS, Wong MCM. Development and validation of the health belief model scale for early childhood caries prevention behaviors of parents. BMC Oral Health. 2025 Jul 2;25(1):1051. doi: 10.1186/s12903-025-06416-1. PMID 40604716
- [Derived] Wang K, Lee GHM, Liu P, Gao X, Wong SYS, Wong MCM. Health belief model for empowering parental toothbrushing and sugar intake control in reducing early childhood caries among young children-study protocol for a cluster randomized controlled trial. Trials. 2022 Apr 12;23(1):298. doi: 10.1186/s13063-022-06208-w. PMID 35413872